CLINICAL TRIAL: NCT01944280
Title: Investigating the Effectiveness of Intradialytic Massage on Cramping in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Sullivan (Other)
Responsible Party: Sponsor-Investigator, Catherine Sullivan, Center Manager, Research, MetroHealth Medical Center
Organization: MetroHealth Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB12-00843
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): The intervention group will receive a 20 minute massage during each hemodialysis treatment for 2 weeks. Most patients receive dialysis 3 times per week resulting in 6 massage sessions. The massage will include both feet and legs up to and including the knee. Massage will include general light centripetal friction and point compression to bellies and myotendinous junction of muscles of the foot and calf not to exceed a perceived pain of 6 on a scale of 1 to 10, 10 being most severe and 1 being no pain.
  Interventions: Other: massage
- control (No Intervention): usual care

INTERVENTIONS:
Other: massage
  Arms: intervention

SUMMARY:
Primary Aim. The primary aim is to determine the effectiveness of intradialytic massage on the frequency and severity of cramping among hemodialysis patients prone to lower extremity cramping during treatment.

Hypothesis: Compared to control patients, intervention patients will be significantly less likely to have intradialytic cramping that requires staff intervention or treatment termination.

This is a study involving 32 (16 intervention, 16 control) hemodialysis patients with frequent lower extremity cramps during treatment. Frequent cramping during dialysis treatments is defined as 1 or more episodes of lower extremity cramps during or after dialysis over the previous 2 weeks. Cramping frequency will be determined by chart notes. Muscle cramping is defined as contraction of the large muscle group of the lower extremities sufficiently painful to require intervention by the dialysis staff for relief.

The intervention group will receive a 20 minute massage of the lower extremities by a trained and licensed massage therapist during each treatment (3x per week) for 2 weeks. The control group will receive usual care by dialysis center staff.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age and <90 years of age.
* On hemodialysis greater than 6 months.
* A stable dry weight for the previous month.
* Frequent cramping during dialysis treatments defined as 1 or more episodes of lower extremity cramps during or after dialysis over the previous 2 weeks.
* Ability to give informed consent.

Exclusion Criteria:

* Sores or wounds on feet or lower legs.
* Dermatitis of lower legs or feet.
* Edema greater than 2+.
* Known history of Deep Vein Thrombosis.
* Vascular access (arteriovenous (A-V) graft, A-V fistula or catheter) for hemodialysis is located in the lower extremity.
* Evidence of open leg wounds, history of lower extremity amputation or documented history of peripheral vascular disease.
* Acute hemodynamic or clinical instability per the dialysis nurse or tech just prior to the intervention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary aim is to determine the effectiveness of intradialytic massage on the frequency and severity of cramping among hemodialysis patients prone to lower extremity cramping during treatment. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashwini Sehgal, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Centers For Dialysis Care, Cleveland, Ohio, United States